CLINICAL TRIAL: NCT03760549
Title: Extension Study for Study ALT-103-201: One-year Follow-up for the 1×10(11th) vp NasoVAX Group
Brief Title: Study of the Safety and Immunogenicity of NasoVAX Extension
Status: Completed | Type: Observational
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALT103-201EXT
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extension of NasoVAX high dose: A serum sample will be collected from each eligible subject who received NasoVAX at the 1×10(11th) vp dose in Study ALT-103-201 for evaluation of influenza hemagglutination assay against influenza A/California/07/2009(H1N1), a strain homologous to the one used for NasoVAX (monovalent AdcoCA09.HA). Ad5 antibody neutralization assay may also be performed.
  Interventions: Drug: Subjects were administered NasoVAX high dose

INTERVENTIONS:
Drug: Subjects were administered NasoVAX high dose — NasoVAX administered by intranasal spray at a single dose of 1×10(11th) viral particles (vp) versus placebo

SUMMARY:
This study is an extension to Study ALT-103-201, a Phase 2a, randomized, double-blind, placebo-controlled trial to evaluate the safety and immunogenicity of NasoVAX in healthy adults 18 to 49 years of age.

DETAILED DESCRIPTION:
This study is an extension to Study ALT-103-201 to evaluate immunogenicity of NasoVAX administered by intranasal spray at a single dose of 1×1011 vp at Day 366 (± 60 days). Up to 15 subjects who received NasoVAX at the 1×10(11th) vp dose in Study ALT-103-201 will be screened, and a serum sample will be collected from each eligible subject for evaluation of influenza HAI assay against influenza A/California/07/2009(H1N1), a strain homologous to the one used for NasoVAX (monovalent AdcoCA09.HA). Ad5 antibody neutralization assay may also be performed.

ELIGIBILITY:
Inclusion:

1. Receipt of NasoVAX at the 1×10(11th) vp dose in Study ALT-103-201
2. Adequate venous access for phlebotomy
3. Provision of written informed consent

Exclusion:

1. Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with the subject providing an adequate blood sample or the subject's ability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All subjects who were previously randomized to the 1×10(11th) vp NasoVAX group in Study ALT-103-201
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Immune response to NasoVAX when administered by intranasal spray at a single dose of 1×10(11th) vp after approximately 1year | Day 366
  Antibody level measured by hemagglutination inhibition titer

SECONDARY OUTCOMES:
Persistence of antivector immune response following NasoVAX administered by intranasal spray at a single 1×10(11th) vp dose after approximately 1year | Day 366
  Antibody level measured by Adenovirus serotype 5 neutralization

CONTACTS AND LOCATIONS:
Overall Officials: Peta-Gay Jackson-Booth, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Optimal Health Research, Rockville, Maryland, United States